CLINICAL TRIAL: NCT02691065
Title: Effect of a Treatment Switch from Protease Inhibitor to Raltegravir-based ART on Myeloid Cell Inflammation in HIV-infected Patients.
Brief Title: Protease Inhibitor Vs. Raltegravir-based ART and Inflammation in HIV Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Jean-Pierre Routy, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-579-MUHC
Record Dates: First submitted 2016-02-17; First posted 2016-02-25 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: HIV
MeSH Terms: interventions — Integrase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrase Inhibitor (Experimental): Switch from protease inhibitor-based regimen to raltegravir-based regimen
  Interventions: Drug: Integrase Inhibitor
- Protease inhibitor (No Intervention): Continuation of protease-inhibitor based regimen

INTERVENTIONS:
Drug: Integrase Inhibitor — Raltegravir
  Arms: Integrase Inhibitor

SUMMARY:
Human immunodeficiency virus (HIV) infection damages body defence mainly by affecting two important white blood cells called cluster of differentiation (CD4) T cells and monocytes. This immune dysfunction leads to persistent inflammation, which is partially resolved with long-term anti-HIV therapy. Importantly, such inflammation increases risk for cardiovascular, diabetes, and kidney diseases. The causes of this inflammation are largely unknown and include HIV itself, presence of other infections, lifestyle characteristics like increased cholesterol levels, obesity, smoking and alcohol abuse. In addition, inflammation can be driven by certain type of anti-HIV therapy called protease inhibitor (PI). PI has been associated with an increase of cholesterol and may contribute to inflammation. A new class of medication that is now available in Canada called integrase inhibitor (II) may have a lesser or no effect on cholesterol levels. Therefore, it is important to study the effect of II on cholesterol levels and inflammation.

The purpose of this study is to assess the inflammatory changes, in the blood of persons treated with PI that will switch to the II or may remain on their PI-containing regimen. By comparing persons continuing their current PI-based regimen with those who switch to II-based regimen, we will know if the change from PI to raltegravir (Isentress), a type of II, decreases lipids and inflammatory markers.

The adult persons living with HIV, who are on PI-based therapy for more than a year, with any CD4 T cell count and plasma viral load below level of detection, will be invited to participate in the study. 40 study participants will be selected by randomization (like a toss of a coin) to either continue PI-based regimen (20 participants) or switch to raltegravir-based regimen (20 participants) for a period of 12 months. Blood samples of the study participants will be drawn before, during and at the end of study to evaluate changes in markers of inflammation, cholesterol level and CD4 T cell and monocyte function. No experimental anti-HIV medication will be used; change of therapy will include raltegravir which is one of currently recommended medications to treat HIV in Canada.

This study will be able to answer this important question whether inflammation can be decreased by switching therapy from PI-based therapy to raltegravir-based therapy. Ultimately, information provided by this study will contribute to the health of persons living with HIV.

ELIGIBILITY:
Inclusion Criteria

1. HIV-1 infected male or female adults greater than or equal to 18 years of age
2. Participants who are on protease-inhibitor-based ART for more than a year
3. Participants with any CD4 T-cell count.
4. Participants with plasma viral load below level of detection (40 copies/mL)
5. Able to understand and sign the informed consent form prior to screening
6. Women of child-bearing potential must have a negative pregnancy test at screening and at Day 1 and agree to use the following approved methods of birth control while on study:

   * Double barrier method (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide);
   * Any intrauterine device (IUD) with published data showing that the expected failure rate is <1% per year (not all IUDs meet this criterion);
   * Male partner sterilization confirmed prior to the female subject's entry into the study; this male is the sole partner for that subject;
   * Approved hormonal contraception;
   * Any other method with published data showing that the expected failure rate is <1% per year.

   Any contraception method must be used consistently, in accordance with the approved product label, and for at least 2 weeks after discontinuation of metformin.
7. Women of non-child-bearing potential as defined as either post-menopausal (12 months of spontaneous amenorrhea and ≥ 45 years of age) or physically incapable of becoming pregnant with documented tubal ligation, hysterectomy or bilateral oophorectomy.
8. Men who are using at least one barrier method of contraception (e.g. condom).

Exclusion Criteria

1. Individuals with a known hypersensitivity/allergy to the Raltegravir.
2. Individuals who are actively participating in an experimental therapy study or who have received experimental therapy within the last three months.
3. Individuals who are suffering from severe systemic diseases (uncontrolled hypertension, chronic renal failure), or active uncontrolled infections
4. Patients who are currently on any integrase inhibitor-based ART.
5. Individuals with a history of congestive heart failure (NYHA I-IV) or individuals having a cardiac pacemaker
6. Severe liver or kidney disease based on physician evaluation
7. Elevated AST or ALT 3-fold above the upper normal limit
8. Elevated alkaline phosphatase 2-fold above upper normal limit
9. Elevated creatinine (above 150 µmol/l)
10. Current use of oral steroids
11. A systemic infection within the last month
12. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Reduction in the frequency of inflammatory monocytes | 12 months
  Phenotypic assessment of peripheral blood monocytes by flow cytometry to determine the percentage of CD14+ CD16+ monocytes. This will be compared between two arms to determine the effect of Raltegravir-based therapy vs protease inhibitor-based therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Routy, MD; FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Chronic Viral Illness Service, McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenabian MA, Mehraj V, Costiniuk CT, Vyboh K, Kema I, Rollet K, Paulino Ramirez R, Klein MB, Routy JP. Influence of Hepatitis C Virus Sustained Virological Response on Immunosuppressive Tryptophan Catabolism in ART-Treated HIV/HCV Coinfected Patients. J Acquir Immune Defic Syndr. 2016 Mar 1;71(3):254-62. doi: 10.1097/QAI.0000000000000859. PMID 26436613
- [Background] Jenabian MA, El-Far M, Vyboh K, Kema I, Costiniuk CT, Thomas R, Baril JG, LeBlanc R, Kanagaratham C, Radzioch D, Allam O, Ahmad A, Lebouche B, Tremblay C, Ancuta P, Routy JP; Montreal Primary infection and Slow Progressor Study Groups. Immunosuppressive Tryptophan Catabolism and Gut Mucosal Dysfunction Following Early HIV Infection. J Infect Dis. 2015 Aug 1;212(3):355-66. doi: 10.1093/infdis/jiv037. Epub 2015 Jan 23. PMID 25616404
- [Background] Mehraj V, Jenabian MA, Vyboh K, Routy JP. Immune Suppression by Myeloid Cells in HIV Infection: New Targets for Immunotherapy. Open AIDS J. 2014 Dec 29;8:66-78. doi: 10.2174/1874613601408010066. eCollection 2014. PMID 25624956
- [Background] Cao W, Mehraj V, Trottier B, Baril JG, Leblanc R, Lebouche B, Cox J, Tremblay C, Lu W, Singer J, Li T, Routy JP; Montreal Primary HIV Infection Study Group; Vezina S, Charest L, Milne M, Huchet E, Lavoie S, Friedman J, Duchastel M, Villielm F, Cote P, Potter M, Lessard B, Charron MA, Dufresne S, Turgeon ME, Rouleau D, Labrecque L, Fortin C, de Pokomandy A, Hal-Gagne V, Munoz M, Deligne B, Martel-Laferriere V, Gilmore N, Fletcher M, Szabo J. Early Initiation Rather Than Prolonged Duration of Antiretroviral Therapy in HIV Infection Contributes to the Normalization of CD8 T-Cell Counts. Clin Infect Dis. 2016 Jan 15;62(2):250-257. doi: 10.1093/cid/civ809. Epub 2015 Sep 8. PMID 26349551
- [Background] Aounallah M, Dagenais-Lussier X, El-Far M, Mehraj V, Jenabian MA, Routy JP, van Grevenynghe J. Current topics in HIV pathogenesis, part 2: Inflammation drives a Warburg-like effect on the metabolism of HIV-infected subjects. Cytokine Growth Factor Rev. 2016 Apr;28:1-10. doi: 10.1016/j.cytogfr.2016.01.001. Epub 2016 Jan 27. PMID 26851985
- [Background] Routy JP, Angel JB, Patel M, Kanagaratham C, Radzioch D, Kema I, Gilmore N, Ancuta P, Singer J, Jenabian MA. Assessment of chloroquine as a modulator of immune activation to improve CD4 recovery in immune nonresponding HIV-infected patients receiving antiretroviral therapy. HIV Med. 2015 Jan;16(1):48-56. doi: 10.1111/hiv.12171. Epub 2014 Jun 2. PMID 24889179